CLINICAL TRIAL: NCT03836807
Title: A Multicenter, Double Blind, Randomised, Parallel Study to Assess Efficacy and Tolerability After Single Administration of Ketoprofen Lysine Salt 40 mg Granules vs Placebo in Subjects With Acute Pain Syndrome After Removal of Molar Teeth
Brief Title: A Study to Assess Efficacy and Tolerability of Ketoprofen 40 mg Granules vs Placebo
Acronym: KSL0117
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSL0117
Record Dates: First submitted 2019-01-28; First posted 2019-02-11 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Acute Pain
Keywords: dental pain; neuralgia
MeSH Terms: conditions — Acute Pain; Toothache; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The double-blinding is provided by Placebo that is identical to OKITASK® 40 mg granules.
  The drug will be packaged and labeled in a manner that will exclude unblinding. IWRS will assign the study drug kit number that should be administrated by the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OKITASK® (Experimental): Single oral administration of Ketoprofen lysine salt 40 mg granules
  Interventions: Drug: OKITASK®
- Placebo (Placebo Comparator): Single oral administration of placebo matching granules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OKITASK® — A single oral dose of OKITASK® 40 mg was administered to patients within 3 hours after extraction of a molar tooth (VAS ≥ 30 mm). Each patient received one sachet that contained KLS 40 mg (equivalent to 25 mg of ketoprofen). The content of the entire sachet was placed on the patient's tongue and swallowed. A glass of water was immediately administered after the intake of the study drug in order to rinse mouth for all subjects.
  Other Names: ketoprofen lysine salt (KLS)
  Arms: OKITASK®
Other: Placebo — A single oral dose of matching Placebo was administered to patients within 3 hours after extraction of a molar tooth (VAS ≥ 30 mm). Each patient received one sachet that contained Placebo. The content of the entire sachet was placed on the patient's tongue and swallowed. A glass of water was immediately administered after the intake of the study drug in order to rinse mouth for all subjects.
  Other Names: Control
  Arms: Placebo

SUMMARY:
Primary objective:

To assess the efficacy of OKITASK® 40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth by comparing AUC0-6h of posttreatment pain profile measured by VAS.

Secondary objectives:

To assess the following efficacy and safety parameters of OKITASK® 40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth:

* Time profile of pain and time profile of pain relief using VAS scales
* Time to first perceptible pain relief (TFPR) and time to meaningful pain relief (TMPR)
* Proportion of patients requiring rescue medication (analgesia) and time to rescue analgesia
* Patient's overall assessment
* Rate of adverse events (AE)

DETAILED DESCRIPTION:
This is a multicenter, double blind, randomized, parallel groups study to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome after removal of a molar tooth.

The patients are assigned to one of two treatment group in 1:1 ratio:

* Group 1. OKITASK® 40 mg - 35 patients;
* Group 2. Placebo - 35 patients. The study was conducted at 3 Russian sites. A total number of enrolled subjects was 70 (35 per each group). Patients' enrollment was competitive.

The study consisted of three periods: screening, study treatment and follow-up. The duration of participation of each subject in the study was to be up to 7±1 days and included: screening (up to 4 days), tooth extraction, randomization and study treatment (1 day), and follow-up (2 days).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Male and female, from 18 years to 65 years (inclusively);
3. Subjects who undergo removal of a non-impacted molar tooth within 3 hours before randomization in the study;
4. Subjects in generally good health (based upon criteria for safe administration of outpatient conscious sedation);
5. Subjects requesting relief for postoperative pain within 3 h after the tooth extraction (VAS ≥30 mm);
6. Subjects willing to undergo observation period for up to 9 hours after the tooth extraction;
7. Ability to complete a 100 mm VAS and a category scale during the observation period (about 9 hours);
8. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study;
9. Contraception (for females): females of child-bearing potential must be using at least one reliable method of contraception, as follows:

   1. hormonal oral, implantable, transdermal, or injectable contraceptives;
   2. a non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide; or should have:
   3. a male sexual partner who agrees to use a male condom with spermicide;
   4. a sterile sexual partner.

Exclusion Criteria:

1. Subjects undergoing extraction of impacted and dystopic teeth, tooth preserving operations, apically positioning flap/vestibuloplasty with free gingival graft from the palate;
2. Subjects undergoing more than one tooth extraction in the same extraction procedure;
3. Subjects undergoing dental implantation simultaneously with tooth extraction;
4. Allergy: ascertained or presumptive hypersensitivity to the active substances (ketoprofen and paracetamol as rescue medication) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to NSAIDs) or allergic reactions in general, which the Investigator considers may affect the outcome of the study;
5. Diseases: relevant history of renal, hepatic, cardiovascular, respiratory (including asthma), skin, haematological, endocrine, gastro-enteric and genitourinary tract or neurological and autoimmune diseases, that may interfere with the aim of the study;
6. Medications: non-steroidal anti-inflammatory drugs (NSAIDS) and other analgesics [in particular ketoprofen, paracetamol and acetylsalicylic acid (ASA)], antihistamines, sedating medications, including herbal and BASs, taken 48 h before surgery;
7. Investigational drug trials: participation in the evaluation of any drug within 3 months before screening (including the last study procedure);
8. Relevant history of drug and alcohol abuse.
9. Positive Pregnancy test in female patients of childbearing potential (including patients in post-menopausal status for less than 2 years).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Lanata, MD, Study Director — Dompé SpA Milan
Locations (3):
- Russia (3):
  - LLC "Centre for Interdisciplinary Dentistry and Neurology", Moscow
  - Federal State Educational Institution "Moscow State Medical Dental University named after Yevdokimov "of the Russian Federation Ministry of Health, Moscow
  - State Autonomous Healthcare Institution of Yaroslavl Region "Clinical Hospital of Emergency care n.a. N.V. Solovyev", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 73 screened patients in the study. 70 of them were randomized into the OKITASK® or Placebo groups by 35 patients per each group.
Groups:
- OKITASK®: Single oral administration of Ketoprofen lysine salt 40 mg granules
  Ketoprofen: 40 mg KLS granules (corresponding to 25 mg ketoprofen)
- Placebo: Single oral administration of placebo granules
  Placebo: 0 mg KLS granules
Period: Overall Study
Arm/Group | OKITASK® | Placebo
Started | 35 | 35
Intent To Treat (ITT) | 35 | 35
Per Protocol (PP) | 33 | 35
Safety Population (SAF) | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: included all randomized patients who received at least one dose of study medication and have at least one post-baseline18 efficacy measurement.
Groups:
- Ketoprofen: Single oral administration of Ketoprofen lysine salt 40 mg granules
  Ketoprofen: 40 mg KLS granules (corresponding to 25 mg ketoprofen)
- Total: Total of all reporting groups
Arm/Group | Ketoprofen | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: AUC0-6h of Pain Intensity Between Time 0 (Baseline Value of VAS) and 6 Hours Post-treatment in the ITT Population.
Description: The primary efficacy endpoint is the pain intensity assessment during 6 hours after molar tooth extraction measured as an area under the curve (AUC) of pain intensity assessed with a visual analogue scale (VAS). More precisely, pain is assessed by a horizontal 100 mm scale where 0 mm = no pain and 100 mm = worst pain imaginable, at the timepoints specified here under in the interval from time 0 (baseline value of VAS) to 6 hours after the drug administration. The AUC0-6h is calculated using the trapezoidal rule. Please note that at 0' (just before taking the first medication) VAS should be >30 mm.
  The higher the score, the worse the result.
Time Frame: time 0', 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-treatment
Population: The Intent-to-treat (ITT) population included all randomized patients who received at least one dose of study medication and have at least one post-baseline18 efficacy measurement; one patient in the ketoprofen group had missing data of the pain intensity VAS and such data were not replaced according to rules for LOCF; hence no AUC for this patient was calculated.
Measure: Mean (Standard Deviation); unit: mm*min
Groups:
- OKITASK: Single oral administration of Ketoprofen lysine salt 40 mg granules
  Ketoprofen: 40 mg KLS granules (corresponding to 25 mg ketoprofen)
Arm/Group | OKITASK | Placebo
Number analyzed (Participants) | 34 | 35
mm*min | 5031 (3250) | 7593 (5402)
Statistical Analysis 1: Comparison: OKITASK vs Placebo; Test type: Superiority; p = 0.020, ANOVA

2. Primary Outcome: AUC0-6h of Pain Intensity Between Time 0 (Baseline Value of VAS) and 6 Hours Post-treatment in the PP Population.
Description: The primary efficacy endpoint is the pain intensity assessment during 6 hours after molar tooth extraction measured as an area under the curve (AUC) of pain intensity assessed with a visual analogue scale (VAS). More precisely, pain is assessed by a horizontal 100 mm scale where 0 = no pain and 100 = worst pain imaginable, at the timepoints specified here under in the interval from time 0 (baseline value of VAS) to 6 hours after the drug administration. The AUC0-6h is calculated using the trapezoidal rule. Please note that at 0' (just before taking the first medication) VAS should be >30 mm.
  The higher the score, the worse the result.
Time Frame: as for outcome 1
Population: The Per protocol population included those patients who had completed the study treatment period, had all assessments for the primary efficacy analysis and considered compliant. The patients were compliant if they did not have any major protocol violations in the course of the study. For the PP population no data could be missing, hence there were no LOCF or other methods applied.
Measure: Mean (Standard Deviation); unit: mm*min
Arm/Group | OKITASK | Placebo
Number analyzed (Participants) | 33 | 35
mm*min | 5099 (3275) | 7593 (5402)
Statistical Analysis 1: Comparison: OKITASK vs Placebo; Test type: Superiority; p = 0.026, ANOVA

3. Secondary Outcome: Time Profile of Pain Intensity Using VAS Scale
Description: This outcome analyzed the evolution and the profile of pain by a horizontal 100 mm Visual Analogue Scale (VAS): 0 no pain - 100 worst pain imaginable at 0' (just before taking the first medication VAS should be >30 mm) and 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240'(4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration. The higher the score, the worse the result.
Time Frame: From time 0 (baseline value of VAS) to 6 hours post-treatment at: 0', 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 35 | 35
mm
  0 min | 45.3 (12.0) | 45.5 (9.9)
  5min | 45.2 (14.2) | 43.9 (11.5)
  10min | 40.4 (16.3) | 40.7 (13.5)
  15min | 34.9 (18.8) | 37.0 (15.5)
  30min | 22.4 (17.9) | 30.9 (17.8)
  45min | 16.2 (16.9) | 24.6 (17.4)
  1h | 13.4 (14.0) | 22.4 (18.0)
  1,5h | 12.1 (12.6) | 22.6 (19.3)
  2h | 11.5 (13.8) | 20.8 (18.1)
  3h | 12.7 (15.6) | 18.2 (18.3)
  4h | 13.6 (13.9) | 18.4 (19.4)
  5h: number analyzed (Participants) | 34 | 35
  5h | 11.8 (9.5) | 16.7 (16.8)
  6h: number analyzed (Participants) | 34 | 35
  6h | 12.6 (9.9) | 16.5 (18.2)
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; at Baseline (at 0'); Test type: Superiority; p = 0.914, ANOVA; The ANOVA model included fixed effect terms for clinical site, time point and treatment. Time point was specified as a repeated measurement; adjusted least square mean = -0.3, 95% CI 2-sided [-5.5 to 5.0]
Statistical Analysis 2: Comparison: OKITASK® vs Placebo; at 5'; Test type: Superiority; p = 0.685, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 1.3, 95% CI 2-sided [-4.9 to 7.4]
Statistical Analysis 3: Comparison: OKITASK® vs Placebo; at 10'; Test type: Superiority; p = 0.930, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -0.3, 95% CI 2-sided [-7.4 to 6.8]
Statistical Analysis 4: Comparison: OKITASK® vs Placebo; at 15'; Test type: Superiority; p = 0.615, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -2.1, 95% CI 2-sided [-10.3 to 6.1]
Statistical Analysis 5: Comparison: OKITASK® vs Placebo; at 30'; Test type: Superiority; p = 0.051, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -8.5, 95% CI 2-sided [-17.0 to 0]
Statistical Analysis 6: Comparison: OKITASK® vs Placebo; at 45'; Test type: Superiority; p = 0.043, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -8.4, 95% CI 2-sided [-16.6 to -0.3]
Statistical Analysis 7: Comparison: OKITASK® vs Placebo; at 1h; Test type: Superiority; p = 0.023, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -9.0, 95% CI 2-sided [-16.7 to -1.3]
Statistical Analysis 8: Comparison: OKITASK® vs Placebo; at 1.5h; Test type: Superiority; p = 0.009, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -10.5, 95% CI 2-sided [-18.2 to -2.7]
Statistical Analysis 9: Comparison: OKITASK® vs Placebo; at 2h; Test type: Superiority; p = 0.018, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -9.3, 95% CI 2-sided [-17.0 to -1.7]
Statistical Analysis 10: Comparison: OKITASK® vs Placebo; at 3h; Test type: Superiority; p = 0.182, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -5.5, 95% CI 2-sided [-13.6 to 2.6]
Statistical Analysis 11: Comparison: OKITASK® vs Placebo; at 4h; Test type: Superiority; p = 0.236, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -4.8, 95% CI 2-sided [-12.9 to 3.2]
Statistical Analysis 12: Comparison: OKITASK® vs Placebo; at 5h; Test type: Superiority; p = 0.320, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -3.6, 95% CI 2-sided [-10.6 to 3.5]
Statistical Analysis 13: Comparison: OKITASK® vs Placebo; at 6h; Test type: Superiority; p = 0.572, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = -2.2, 95% CI 2-sided [-10.0 to 5.6]

4. Secondary Outcome: Time Profile of Pain Relief Using VAS Scale
Description: This outcome analyzed the evolution of pain relief after administration of OKITASK® and after administration of Placebo, assessed by a horizontal 100 mm Visual Analogue Scale (VAS): 0 no pain relief - 100 maximum relief imaginable at: 0' (just before taking the first medication VAS should be >30 mm) and 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240'(4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration. The higher the score, the best the result.
Time Frame: From time 0 (baseline value of VAS) to 6 hours post-treatment at: 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 35 | 35
mm
  at 5' | 12.7 (14.0) | 10.1 (9.7)
  at 10' | 20.3 (18.8) | 16.0 (14.6)
  at 15' | 31.6 (25.3) | 22.7 (20.5)
  at 30' | 57.6 (31.4) | 35.2 (29.3)
  at 45' | 68.9 (30.9) | 47.8 (34.2)
  at 1h | 73.5 (29.3) | 54.9 (34.9)
  at 1.5h | 79.7 (24.7) | 57.4 (35.6)
  at 2h | 82.1 (21.3) | 60.1 (35.9)
  at 3h | 82.8 (19.7) | 66.1 (34.2)
  at 4h | 80.5 (23.5) | 69.7 (30.8)
  at 5h | 81.4 (21.8) | 73.9 (25.0)
  at 6h | 79.8 (22.7) | 75.8 (25.4)
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; at 5'; Test type: Superiority; p = 0.361, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 2.7, 95% CI 2-sided [-3.1 to 8.4]
Statistical Analysis 2: Comparison: OKITASK® vs Placebo; at 10'; Test type: Superiority; p = 0.298, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 4.2, 95% CI 2-sided [-3.8 to 12.3]
Statistical Analysis 3: Comparison: OKITASK® vs Placebo; at 15'; Test type: Superiority; p = 0.112, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 8.9, 95% CI 2-sided [-2.1 to 19.8]
Statistical Analysis 4: Comparison: OKITASK® vs Placebo; at 30'; Test type: Superiority; p = 0.003, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 22.3, 95% CI 2-sided [7.8 to 36.8]
Statistical Analysis 5: Comparison: OKITASK® vs Placebo; at 45'; Test type: Superiority; p = 0.008, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 21.2, 95% CI 2-sided [5.6 to 36.7]
Statistical Analysis 6: Comparison: OKITASK® vs Placebo; at 1h; Test type: Superiority; p = 0.018, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 18.7, 95% CI 2-sided [3.3 to 34.0]
Statistical Analysis 7: Comparison: OKITASK® vs Placebo; at 1.5h; Test type: Superiority; p = 0.003, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 22.3, 95% CI 2-sided [7.7 to 37.0]
Statistical Analysis 8: Comparison: OKITASK® vs Placebo; at 2h; Test type: Superiority; p = 0.003, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 22.0, 95% CI 2-sided [8.0 to 36.1]
Statistical Analysis 9: Comparison: OKITASK® vs Placebo; at 3h; Test type: Superiority; p = 0.015, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 16.7, 95% CI 2-sided [3.4 to 30.0]
Statistical Analysis 10: Comparison: OKITASK® vs Placebo; at 4h; Test type: Superiority; p = 0.103, ANOVA; adjusted least square mean = 10.8, 95% CI 2-sided [-2.2 to 23.9]
Statistical Analysis 11: Comparison: OKITASK® vs Placebo; at 5'; Test type: Superiority; p = 0.311, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 5.9, 95% CI 2-sided [-5.6 to 17.5]
Statistical Analysis 12: Comparison: OKITASK® vs Placebo; at 6h; Test type: Superiority; p = 0.638, ANOVA; [statistical method as in outcome 3, analysis 1]; adjusted least square mean = 2.8, 95% CI 2-sided [-9.0 to 14.5]

5. Secondary Outcome: AUC5min-6h of Pain Relief Profile in the ITT and in the PP Populations
Description: In addition, area under the curve for pain relief assessment since 5 minutes till 6 hours after the drug administration was evaluated.
Time Frame: from 5 min to 6 hours post-dose
Population: ITT population included all randomized patients who received at least one dose of study medication and have at least one post-baseline 18 efficacy measurement; one patient in the ketoprofen group had missing data of the pain intensity VAS and such data were not replaced according to rules for LOCF; hence no AUC for this patient was calculated.
  PP population included those patients who had completed the study treatment period, had all assessments for the primary efficacy analysis and compliant.
Measure: Mean (Standard Deviation); unit: mm*min
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 34 | 35
mm*min
  ITT population | 27445 (6456) | 22103 (9209)
  PP population: number analyzed (Participants) | 33 | 35
  PP population | 27362 (6538) | 22103 (9209)
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; in the ITT population; Test type: Superiority; p = 0.007, ANOVA
Statistical Analysis 2: Comparison: OKITASK® vs Placebo; in the PP population; Test type: Superiority; p = 0.009, ANOVA

6. Secondary Outcome: Time to First Perceptible Relief (TFPR)
Description: TFPR was measured by stopwatches, a timepiece designed to measure the amount of time that elapses between its activation and deactivation. Upon study drug administration the patients immediately started a stopwatch, once the patient felt first perceptible pain relief, the stopwatch was stopped.
  The time between activation and deactivation of a stopwatch defined the outcome measure data. The shortest the time, the better the outcome.
  Kaplan-Meier estimation of TFPR was expressed by median and 95% CI.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 35 | 35
minutes | 18.5 [13.6 to 24.1] | 31.4 [22.0 to 43.0]
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; Test type: Superiority; p = 0.004, Log Rank

7. Secondary Outcome: Time to Meaningful Pain Relief (TMPR)
Description: TMPR will be measured by stopwatches, a timepiece designed to measure the amount of time that elapses between its activation and deactivation. Upon study drug administration the patients will immediately start a stopwatch, once the patient feels meaningful perceptible pain relief, the stopwatch is stopped.
  The time between activation and deactivation of a stopwatch defines the outcome measure data.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 35 | 35
Minutes | 36.9 [26.9 to 42.4] | 58.4 [41.9 to 129.8]
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; Test type: Superiority; p = 0.002, Log Rank

8. Secondary Outcome: Number of Participants With an Overall Assessment Score of "Very Good", "Satisfactory", "Poor" or "Very Poor" on a (Patient's Overall Assessment) on a 5-point Scale
Description: The patients were asked to provide their current overall assessment answering the question "Considering all the ways that the pain affects you, how well are you doing? The patients marked the answer on the 5-point scale: 1 = very good, 2 = good, 3= satisfactory, 4 = poor, 5 = very poor.
  If a patient takes rescue medication, the Patient's overall assessment will be performed after the last VAS assessment.
Time Frame: Day 1 at 360' or > 60' in case of early discontinuation.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | OKITASK® | Placebo
Number analyzed (Participants) | 35 | 35
participants
  Very good | 6 | 2
  good | 22 | 24
  Satisfactory | 7 | 9
  poor | 0 | 0
  no data | 0 | 0
Statistical Analysis 1: Comparison: OKITASK® vs Placebo; Test type: Superiority; p = 0.480, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From screening day (-4) to follow up ( day 3 +/- 1), up to day 3 post-dose.
Description: More specifically, adverse events are assessed at:
  * Screening days (day -4 to day 1)
  * Baseline ( day 1, pre-dose)
  * following time post-dose: 0.08h; 0.17h; 0.25h; 0.5h; 0.75h; 1h; 1.5h; 2h; 3h; 4h; 5h; 6h.
  * day one
  * follow-up ( day 3 +/- 1)
Arm/Group | OKITASK® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 1/35
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OKITASK® (N=35) | Placebo (N=35)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03836807/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03836807/SAP_001.pdf